CLINICAL TRIAL: NCT05560295
Title: Fertility-enhancing Hysteroscopic Surgery; Multi-center Retrospective Cross-sectional Study of Reproductive Outcome
Brief Title: Hysteroscopic Surgery; Retrospective Cross-sectional Study of Reproductive Outcome
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Associate Professor, University of Jordan
Other Study IDs: Hysteroscopic surgery
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Hysteroscopic Metroplasty and Myomectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Naser Al-Husban — uterine surgery

SUMMARY:
study of the effect of hysteroscopic sptoplast and hysteroscopic myomectomy on reproductive performance of patients with infertility and /or miscarriages

DETAILED DESCRIPTION:
Retrospective study and analysis of the reproductive outcome in patients who underwent hysteroscopic surgery for infertility at Jordan university hospital and Al-Noor fertility centre in Amman, Jordan in the period September 2016-october 2021. Patients were followed up for a minimum of 6 months after surgery. Resection of uterine septum or submucosal fibroids were included. Data was obtained from the electronic and paper-based clinical files for patients who were operated upon at these hospitals. Patients who missed follow up after the operation will be contacted by phone or invite them for a clinic review to know of their fertility status and pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* those with primary or secondary infertility of more than 1 year with normal seminal fluid analysis, normal female hormonal profile, patent fallopian tubes bilaterally (as confirmed by hysterosalpingography HSG), normal thyroid function, no previous uterine surgery and no medical diseases.
* Cases with recurrent miscarriages were those with 2 or more first or second trimester miscarriages of an apparently normal singleton fetus with no hormonal, endocrine or maternal or paternal karyotype abnormalities and with no previous history of term pregnancy(s).

Exclusion Criteria:

* All patients who were operated upon outside the context of infertility (heavy bleeding…etc), patients with combined (maternal and paternal) infertility factors,
* Patients with history of any number of term pregnancy,
* Previous uterine surgery,
* Patients with medical diseases,
* Those with abnormal female hormonal profile,
* Those with other potential factors for infertility including endometriosis
* Patients with incomplete or missing data and could not be contacted.
* Patients who had myomectomy or septal resection done using bipolar hysteroscopy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — infertility patients
Study Population: female population with infertility or recurrent miscarriages who have uterine septum or fibroids
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 6 months
  spontaneous

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Husban N, Odeh O, AlRamahi M, Qadri S, Al-Husban H. Fertility-enhancing hysteroscopic surgery; multi-center retrospective cohort study of reproductive outcome. BMC Womens Health. 2023 Aug 29;23(1):459. doi: 10.1186/s12905-023-02562-2. PMID 37644542